CLINICAL TRIAL: NCT00001377
Title: Familial Prostate Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940041; 94-C-0041
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-12

CONDITIONS: Neoplastic Syndromes, Hereditary; Prostatic Neoplasms
Keywords: Familial; Inherited Prostate Cancer; Linkage; Prostate Cancer
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary; Prostatic Neoplasms

SUMMARY:
The purpose of this study is to identify affected individuals in families with prostate cancer and to use this information to identify genetic markers closely-linked to the disease gene.

DETAILED DESCRIPTION:
The purpose of this study is to identify affected individuals in families with prostate cancer and to use this information to identify genetic markers closely-linked to the disease gene.

ELIGIBILITY:
Families will be identified with two or more first degree relatives affected with prostate cancer or with one male with prostate cancer that developed before age 55.

Must have clinical evidence of prostate cancer in the family.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1993-12; Study Completion 2000-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Vocke CD, Pozzatti RO, Bostwick DG, Florence CD, Jennings SB, Strup SE, Duray PH, Liotta LA, Emmert-Buck MR, Linehan WM. Analysis of 99 microdissected prostate carcinomas reveals a high frequency of allelic loss on chromosome 8p12-21. Cancer Res. 1996 May 15;56(10):2411-6. PMID 8625320
- [Background] Bright RK, Vocke CD, Emmert-Buck MR, Duray PH, Solomon D, Fetsch P, Rhim JS, Linehan WM, Topalian SL. Generation and genetic characterization of immortal human prostate epithelial cell lines derived from primary cancer specimens. Cancer Res. 1997 Mar 1;57(5):995-1002. PMID 9041206
- [Background] Emmert-Buck MR, Vocke CD, Pozzatti RO, Duray PH, Jennings SB, Florence CD, Zhuang Z, Bostwick DG, Liotta LA, Linehan WM. Allelic loss on chromosome 8p12-21 in microdissected prostatic intraepithelial neoplasia. Cancer Res. 1995 Jul 15;55(14):2959-62. PMID 7606709